CLINICAL TRIAL: NCT06791902
Title: Study on Preliminary Safety and Efficacy of Adaptive DBS Aligned to Locomotor States to Improve Locomotor Functions in Parkinson's Patients
Acronym: AdapGAIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jocelyne Bloch (Other)
Responsible Party: Sponsor-Investigator, Jocelyne Bloch, Professor, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AdapGAIT
Record Dates: First submitted 2025-01-09; First posted 2025-01-24 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
Keywords: walking deficits; DBS; Parkinson; gait problems; Deep Brain Stimulation; adaptive DBS; aDBS
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Adaptive DBS (Experimental)
  Interventions: Device: Adaptive DBS

INTERVENTIONS:
Device: Adaptive DBS — Adapting DBS stimulation based on locomotor states to alleviate gait deficits

SUMMARY:
At present, there is no cure for Parkinson's disease. The standard treatment involves taking dopaminergic drugs. When drugs lose their effectiveness, they can be supplemented by Deep Brain Stimulation (DBS) therapy. Medication and deep brain stimulation are effective for motor problems such as tremors, slowness of movement, and muscle stiffness. However, there is no effective treatment for walking and balance problems that occur during the course of the disease.

DBS neurostimulators not only stimulate, but also record brain activity in the region in which the electrodes are implanted. This brain activity changes over time, depending on the individual's general state (i.e., medication, eating), movements (sitting, standing or walking) and motor problems (i.e., problems of gait initiation and termination, balance problems and freezing of gait).

Adaptive deep brain stimulation (aDBS) makes it possible to change the stimulation according to brain activity, and thus to these different states. This method involves using the usual Medtronic Percept neurostimulator with its adaptive therapy active. Additional investigational features for adaptive therapy are available within the study.

In this study, we want to evaluate whether adaptive deep brain stimulation is safe and effective in improving walking problems in people with Parkinson's disease.

DETAILED DESCRIPTION:
The hypotheses of the current study are that:

HYPOTHESIS 1: Adaptive DBS, aligned in time to the occurrence of locomotor states, facilitates gait initiation, termination, turning, symmetry and adaptations to obstacles by titrating the delivery of stimulation to the dynamics of gait.

HYPOTHESIS 2: Enforcing that biomarkers of FoG never exceed an abnormally-high value prevents the occurrence of freezing of gait.

The resulting observations will establish a rigorous understanding of motor state-dependent DBS modulations that will open new avenues for the design of evidence-based DBS strategies for locomotor deficits.

The study is divided into 3 different phases, which will take place on 3 different days at CHUV, and will be spread over a maximum of 5 weeks:

PHASE 1: Eligibility (1 day at CHUV)

* Evaluate Feasibility for aDBS
* Characterize DBS and Movement Modulations
* Assess Global Parkinsonian State

PHASE 2: aDBS therapy setup and efficacy evaluation in different conditions (between 2 to 3 days at CHUV)

* Optimize aDBS Parameters
* Test Safety and Performance
* Evaluate Stability and Robustness
* Daily Life Use of aDBS

The 2 to 3 days of Phase 2 will happenoccur within 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with typical or atypical forms of Parkinson's disease; Suffering from gait or balance disorders;
* Implanted with a full Medtronic Percept suite (neurostimulator Percept PC Model B35200 or Percept RC Model B35300; with bilateral leads (Medtronic Legacy leads (Models 3387 and 3389) or Medtronic SenSightTM Directional Lead (models B33015 and B33005)) and lead extensions (Medtronic extensions (Model 37085 and 37086) or SenSightTM extension (model B34000)), or Medtronic SenSightTM Connector Plug (Model B31061));
* Exhibit modulations in at least one frequency band of the LFP that are related to locomotor states or gait deficits.
* Aged 18 years-old or more;
* Must provide and sign the study's Informed Consent prior to any study-related procedures;
* Able to understand and interact with the study team in French;
* Agree to comply in good faith with all conditions of the recordings, and to attend all required study procedures

Exclusion Criteria:

* Exclusive use of interleaved DBS programs that are incompatible with aDBS;
* High impedances or artefacts in neural signals that obstruct the detection of motor-related biomarkers for adaptive DBS;
* Changes in DBS amplitudes (increase/decrease) not well tolerated;
* Secondary causes of gait problems independent of PD;
* Inability to follow the procedures of the study independently;
* History of major psychiatric disorders or major neurocognitive disorders, as considered by the investigators in according with treating physicians;
* Major changes in PD treatments planned within the course of the study;
* History of drug or alcohol abuse in the past 5 years;
* Pregnancy;
* Participation in another investigational study in the preceding 30 days or during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Through study completion, a maximum of 5 weeks
  Occurrence of adverse events and serious adverse events that are deemed related or possibly related to the study procedures, or the use of the investigational system during the duration of the study

SECONDARY OUTCOMES:
Gait performance | At Phase 1 (Day1) and Phase 2 (2 to 3 days within a maximum of 5 weeks from Day1) of the study.
  Timed up-and-go (TUG) task and 10m walk test are tests used to test used to assess gait speed and sit ro stand and gait ability. In the TUG cognitive the participant is also asked to perform a cognitive task when performing the motor task to see the gait ability during dual-task.
Freezing of Gait occurances | At Phase 1 (Day1) and Phase 2 (2 to 3 days within a maximum of 5 weeks from Day1) of the study.
  - The 360° turn test is used to assess freezing during turn. It measures the time it takes to make a full turn on oneself and the number of steps.
  • A custom-made freezing of gait (FOG) circuit is designed to assess the occurrence of freezing of gait. Participants are asked to perform tasks known to favour freezing of gait occurrence. Participants can use their habitual assistive device and perform the task at comfortable speed.
Global Parkinsonian State | At Phase 1 (Day1) and Phase 2 (2 to 3 days within a maximum of 5 weeks from Day1) of the study.
  The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III scale will be performed to evaluate the general motor state of the participant.18 items, score range: 0 (mild) - 132 (severe)
Changes in neural patterns | At Phase 1 (Day1) and Phase 2 (2 to 3 days within a maximum of 5 weeks from Day1) of the study.
  Evaluation of changes in neural patterns in response to adaptive protocols that are aligned in time to biomarkers of locomotor states / transitions. Measured variables: Changes in neural signals recorded with the implantable system across all the aforementioned locomotor tasks.
Sustained efficacy of adaptive DBS during activities of daily life - kinematics parameters | At Phase 2, during the last day of the study (2nd or 3rd day of Phase 2 within a maximum of 5 weeks from Day1 of Phase 1).
  Out-of-the-lab kinematic monitoring is used to evaluate the evolution of the gait pattern in an ecological environment. Participants will be asked to wear a pair of Nushu X sensorized shoes (Magnes AG, Swizterland - CE-marked as electronic device) with integrated motion feedback sensors during the phase 3 of the study, at CHUV. To monitor the rest of the body kinematics, sensors (Physilog, Mindmaze, Switzerland) will be placed on both wrists of the participants.
Sustained efficacy of adaptive DBS during activities of daily life - questionnaire | At Phase 2, during the last day of the study (2nd or 3rd day of Phase 2 within a maximum of 5 weeks from Day1 of Phase 1).
  Evaluation of aDBS in activities of daily living questionnaire is a self-administered questionnaire designed within the scope of this study. It will evaluate the perceived gait quality, and overall motor performance with aDBS during the day

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No